CLINICAL TRIAL: NCT05399147
Title: Tube First Technique as a Conduit for Easy and Fast Firberoptic Intubation
Brief Title: Tube 1st Technique for Easy Fiberoptic Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amr Gaber, lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: fiberoptic intubation
Record Dates: First submitted 2022-03-19; First posted 2022-06-01 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Difficult Intubation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- classic group (CL group) (Other): 20 patients will be enrolled to be intubated using the classic usual technique
  Interventions: Other: fiberoptic intubation classic technique
- tube 1st group (TF group) (Other): 20 patients will be enrolled to be intubated using the tube 1st technique
  Interventions: Other: fiberoptic intubation tube 1st technique

INTERVENTIONS:
Other: fiberoptic intubation classic technique — classic fiberoptic intubation
  Arms: classic group (CL group)
Other: fiberoptic intubation tube 1st technique — tube 1st technique
  Arms: tube 1st group (TF group)

SUMMARY:
the aim of this work is to study how this technique will make nasal fiberoptic intubation easier and faster than the usual classic technique

DETAILED DESCRIPTION:
Difficult intubation is one of the most significant issues anesthesiologists deal with, occasionally. Among these, mandibulofacial deformities face the biggest challenge in intubation and make an anticipated difficult airway (1), due to short length of mandible (HLM), short thyromental distance (TMD), short inter horizontal -incisors gap (IIG) and high grade modified Mallampati test (MMT) (2).

There are several strategies to approach these patients and each technique has unique benefits that should be used on experience. Sitting endotracheal intubation is a useful technique for airway control, in patients with difficult airway or in patients in whom maintenance of the upright posture is beneficial (3), A difficult airway is defined as difficulty with facemask ventilation, difficulty with tracheal intubation, or both (3). According to new updates on difficult airway management, by the American Society of Anesthesiologists, there are non-invasive and invasive interventions for the management of difficult airway. Non-invasive interventions include, without being limited to: awake intubation, video-assisted laryngoscopy, intubating stylets or tube-changers, supraglottic airway (SGA) for ventilation (e.g., LMA, laryngeal tube), SGA for intubation (e.g., ILMA), rigid laryngoscopic blades of variousdesign and size, fiberoptic-guided intubation, and lighted stylets or light wands, while invasive interventions include surgical or percutaneous airway, jet ventilation and retrograde intubation (4).

Attaching a nasal airway to a breathing circuit as a tool to assist or control ventilation is a very helpful trick to have in challenging airway management situations.

Typically, Fiberoptic bronchoscope is passed through the more patent nostril to follow the major nasal pathway at the floor of the nose along the superior aspect of the hard palate, the lateral aspect of the nasal septum inferior to the lower turbinate to reach the nasopharynx where the operator identifies the pharyngeal structures, such as the base of the tongue and/or the epiglottis that are mostly "in-fall" precluding clear views of the larynx requiring a jaw thrust to visualize the laryngeal structures for patients planned to be intubated under general anesthesia [5,6].

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20 and 60 years,
2. ASA Class I& II,
3. Maxillofacial surgeries ex: mandibular surgery, orthognathic surgery and dental extraction surgery,
4. Other surgeries like: oral graft surgery, facial trauma, limited mouth opening ex: submandibular and facial abscess.

Exclusion Criteria:

1. Patient's refusal,
2. ASA III or more,
3. Intrinsic and idiopathic coagulopathy,
4. known allergy to any of the study medications,
5. furthermore, patients were excluded if they had severe hypoxemias due to sever cardiac or lung disease

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
time 1 | baseline
  time 1 = time from start from start of introducing the bronchoscope till viewing the vocal cord measured in seconds.

SECONDARY OUTCOMES:
other measures | baseline
  1. total dose of propofol during procedure measured in mg

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

REFERENCES:
- [Background] Mak PH, Ooi RG. Submental intubation in a patient with beta-thalassaemia major undergoing elective maxillary and mandibular osteotomies. Br J Anaesth. 2002 Feb;88(2):288-91. doi: 10.1093/bja/88.2.288. PMID 11883389
- [Background] Allahyary E, Ghaemei SR, Azemati S. Comparison of six methods for predicting difficult intubation in obstetric patients. Iran Red Crescent Med J. 2008;10:197-204.
- [Background] Fontanarosa PB, Goldman GE, Polsky SS, Schuckman HA, Poyle M. Sitting oral-tracheal intubation. Ann Emerg Med. 1988 Apr;17(4):336-8. doi: 10.1016/s0196-0644(88)80775-3. PMID 3354936
- [Background] Apfelbaum JL, Hagberg CA, Caplan RA, Blitt CD, Connis RT, Nickinovich DG, Hagberg CA, Caplan RA, Benumof JL, Berry FA, Blitt CD, Bode RH, Cheney FW, Connis RT, Guidry OF, Nickinovich DG, Ovassapian A; American Society of Anesthesiologists Task Force on Management of the Difficult Airway. Practice guidelines for management of the difficult airway: an updated report by the American Society of Anesthesiologists Task Force on Management of the Difficult Airway. Anesthesiology. 2013 Feb;118(2):251-70. doi: 10.1097/ALN.0b013e31827773b2. No abstract available. PMID 23364566
- [Background] Wheeler M, Ovassapian A. Fiberoptic endoscopy-aided techniques. In: Benumof's airway management: principles and practice, 2nd ed., vol. 27(5). Mosby Elsevier Philadelphia; 2010. p. 461-67.
- [Background] Murphy MF. Applied functional anatomy of the airway. In: Manual of emergency airway management, 3rd ed., vol. 3(2). USA: Lippincott Williams & Wilkins; 2008.p. 37-46.